CLINICAL TRIAL: NCT01134731
Title: Paliperidone and Lithium in the Treatment of Suicidality - Treatment Indication and Epigenetic Regulation
Acronym: AFSP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Foundation for Suicide Prevention (Other); Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Dr. Richard Shelton, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F100329001
Record Dates: First submitted 2010-05-20; First posted 2010-06-02 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Major Depressive Disorder; Suicidal Ideation
Keywords: depression; suicidality; Major Depressive Disorder, current episode, with suicidality
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation; Depression | interventions — Paliperidone Palmitate; Lithium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- paliperidone (Experimental): dose escalation , levels 1-5 daily dosing ranged from 1-5mg
  Interventions: Drug: paliperidone
- lithium (Active Comparator): dose escalation, level 1-5 daily dosing 300-1500mg
  Interventions: Drug: lithium
- placebo (Placebo Comparator): 1-5 placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: paliperidone — 1-5 mg daily (QD)
  Arms: paliperidone
Drug: lithium — 300-1500mg QD
  Arms: lithium
Drug: Placebo — 1-5 placebo capsules
  Arms: placebo

SUMMARY:
The study aims to use a combined clinical and translational approach to identify an efficient pharmacotherapy for the acute management of suicidality and the epigenetic regulation associated with the treatment.The primary objective is a clinical trial to compare the efficacy of paliperidone versus lithium and placebo as adjunctive therapy to the standard of care antidepressants in the acute management of suicidality in depressed subjects.

Specific Aims 1 and 2 are described in detail below. Analysis for Specific Aim 2 is still underway.

DETAILED DESCRIPTION:
Specific Aim 1: The atypical antipsychotic, paliperidone, when initiated simultaneously with an antidepressant, is superior to lithium plus antidepressant in the early intervention of suicidality in patients with Major Depressive Disorder (MDD). The goal of this aim is to examine the clinical efficacy of paliperidone in reducing suicidality, with a focus on early intervention. The hypothesis is based on our recently completed pilot study in which we found that the atypical antipsychotic, risperidone, had a rapid onset of action to reduce suicidality in patients with MDD. In view of a shortage in acute pharmacological management of suicidality, this study will provide an important new treatment option for the life threatening psychiatric condition.

Specific Aim 2: Both paliperidone and lithium regulate epigenetics by stabilizing DNA methylation, which is correlated with inhibition of glycogen synthase kinase-3 (GSK3) activity and improved clinical symptoms. This exploratory aim is developed based on the recent findings that DNA methylation is involved in regulation of mood, behavior, and cognition, and the enzyme of this epigenetic mechanism - DNA methyltransferase-1 (DNMT1) is regulated by the therapeutic target Glycogen synthase kinase 3 (GSK3). We will measure the expression of DNMTs and DNA methylation of global DNA, Brain-derived neurotrophic factor (BDNF), and Tropomyosin receptor kinase B (TrkB) in peripheral blood before and after study drug treatment, and analyze their correlation with GSK3 activity and clinical symptoms in response to treatment. Outcomes from this study will provide important new information in future development of more effective treatment options for suicidality targeting epigenetic regulation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects who are able to provide informed consent
2. 19-65 years of age
3. Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) diagnosis of MDD by MINI International Neuropsychiatric Interview (MINI) and confirmed by psychiatric interview
4. Currently experiencing a depressive episode with suicidality (defined as having current suicidal thoughts occurring at least 3 out of 7 days in a week).
5. Montgomery-Asberg Depression Rating Scale (MADRS) must include a total score > 25 and a suicidal sub-score > 4.

Exclusion Criteria:

1. Depressed patients without suicidality, patients with severe psychotic features or with primary diagnoses of bipolar disorder (BD), schizophrenia, schizoaffective disorder, or generalized anxiety disorder (GAD), and subjects who have been taking lithium or an antipsychotic in the past 2 weeks
2. Those with uncontrolled medical illnesses. Participants must be on any new medications for at least 30 days to be considered medically stable.
3. For patients with panic disorder, post-traumatic stress disorder (PTSD), borderline personality disorder (BPD), etc. be sure that MDD is the primary diagnosis. When in doubt, decisions will be made on a case-by-case basis.
4. Pregnant women.
5. Allergic to paliperidone, to any other ingredient in paliperidone ER or paliperidone palmitate, or to risperidone.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Shelton, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were male and female, aged 19- 65 years old, recruited as outpatients from the general public.
Groups:
- Paliperidone: dose escalation, levels 1-5 daily dosing range from 1-5 mg
- Lithium: mood stabilizer
  dose escalation levels 1-5 daily dosing lithium: 300-1500mg daily (QD)
- Placebo: 1-5 capsules
Period: Overall Study
Arm/Group | Paliperidone | Lithium | Placebo
Started | 23 | 21 | 10
Completed | 10 | 10 | 2
Not Completed | 13 | 11 | 8
Not completed — Adverse Event | 3 | 2 | 1
Not completed — Physician Decision | 2 | 2 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 1
Not completed — Lost to Follow-up | 5 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Paliperidone 1-5mg; Lithium 600-1500mg: daily
- Placebo 1-5 Capsules: 12 weeks
- Total: Total of all reporting groups
Arm/Group | Paliperidone 1-5mg | Lithium 600-1500mg | Placebo 1-5 Capsules | Total
Number analyzed (Participants) | 23 | 21 | 10 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 10 | 54
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 10 | 54
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 10 | 54

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of Beck Scale for Suicidal Ideation of Three Treatment Groups (Paliperidone, Lithium and Placebo) After 3 Months of Treatment
Description: The Beck Scale for Suicidal Ideation will be used to measure the efficacy of the study drugs. The primary outcome measure is the Beck Suicide Scale Self Report. The primary outcome measure is the Beck Suicide Scale Self Report. It has 21 questions (subscales) with values ranging from 0-2. Therefore the total score ranges from 0-42, with lower scores indicating better outcomes. The subscales were summed to achieve a total score.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Paliperidone: dose escalation , levels 1-5 daily dosing ranged from 1-5mg
  paliperidone: 1-5 mg qd
- Placebo: placebo comparator, 1-5 capsules
Arm/Group | Paliperidone | Lithium | Placebo
Number analyzed (Participants) | 23 | 21 | 10
units on a scale | 22.1 (8.6) | 22.1 (8.6) | 21.3 (9.6)

2. Secondary Outcome: Mean Score of Montgomery-Asberg Depression Scale of Three Treatment Groups (Paliperidone, Lithium and Placebo) After 3 Months of Treatment
Description: The Montgomery-Asberg Depression Rating Scale will be used to measure depressive symptoms to determine the efficacy of the study drugs. It has 10 items (subscales) ranging from 0-6. Therefore the total score ranges from 0-60, with lower scores indicating better outcomes. The subscales were summed for a total score.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone | Lithium | Placebo
Number analyzed (Participants) | 23 | 21 | 10
units on a scale | 37.5 (5.6) | 39.6 (4.1) | 39.2 (8.1)

ADVERSE EVENTS:
Time Frame: Adverse event reporting started 3/1/2011 and stopped 10/15/2014
Description: The primary outcome variable was the Beck Scale for Suicide Ideation (BSSI, items 1-19).
Arm/Group | Paliperidone | Lithium | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21 | 0/10
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21 | 0/10

LIMITATIONS AND CAVEATS:
The inherent risk of the condition and concerns about the safety of the study, the high risk of impulsive and aggressive behavior, and high levels of distress making placebo-controlled studies difficult. Placebo arm terminated early due to dropout.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less